CLINICAL TRIAL: NCT06234072
Title: Comparison of Neoadjuvant Treatment for Pancreatic Cancer: Astragalus Combined With Gemcitabine Versus Gemcitabine Alone - A Single-Center, Randomized, Double-Blind Study
Brief Title: Comparing Astragalus Plus Gemcitabine to Gemcitabine Alone as Neoadjuvant Treatment for Pancreatic Cancer Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shenzhen University General Hospital (Other)
Responsible Party: Principal Investigator, Xianbin Zhang, Principal Investigator, Shenzhen University General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GEN-SUR-001; 82104596 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Astragalus + Gemcitabine (Experimental): Participants will receive Astragalus in combination with Gemcitabine by intravenous infusion (IV).
  Participants will receive IV infusion of 20ml of Astragalus injection (the content of Astragalus crude drug is 2g/ml plus 250ml of normal saline 1 day before chemotherapy, once a day for 21 consecutive days constitute a course of treatment a total of 4 courses of treatment.
  Gemcitabine is one of the main chemotherapy drugs used to treat pancreatic cancer.
  Interventions: Drug: Astragalus + Gemcitabine
- Gemcitabine alone (Active Comparator): Participants will receive Neoadjuvant Chemotherapy of Gemcitabine 1000 mg/m2 as a 30- to 40-minute infusion (maximum 40 minutes) administered weekly for 7 weeks followed by a week of rest (8-week cycle; cycle 1 only), followed by cycles of weekly administration for 3 weeks (on days 1, 8, and 15) followed by one week of rest (4-week cycle).
  Interventions: Drug: Gemcitabine alone

INTERVENTIONS:
Drug: Astragalus + Gemcitabine — Participants will receive Astragalus combined with Gemcitabine. Astragalus, a traditional Chinese medicine, exhibits promising potential in cancer treatment. Studies suggest its role in regulating immune responses, suppressing tumors, and improving overall treatment outcomes in cancer patients. Astragalus combined with chemotherapeutic drug such as Gemcitabine is a popular complementary and alternative therapy used for cancer patients because it can increase therapeutic effects and decrease side effects. This synergistic approach holds potential for more effective and targeted therapeutic outcomes in pancreatic cancer patients.
  Arms: Astragalus + Gemcitabine
Drug: Gemcitabine alone — Gemcitabine is a potent chemotherapy drug widely employed in treating various cancers, including pancreatic cancer. As a nucleoside analog, it disrupts DNA synthesis, impeding cancer cell proliferation. Gemcitabine is administered intravenously and has shown efficacy in alleviating symptoms, improving survival rates, and enhancing the quality of life for patients undergoing cancer treatment.
  Arms: Gemcitabine alone

SUMMARY:
This study compare the efficacy of Astragalus combined with Gemcitabine to Gemcitabine alone as neoadjuvant treatment for pancreatic cancer.

DETAILED DESCRIPTION:
Astragalus is a commonly used traditional Chinese medicine in China, which has been widely applied to enhance the immunomodulatory function of the body and suppress the growth of tumors. It was often combined with other herbs to strengthen the body against disease. The effects and mechanisms of Astragalus and Shenqi Fuzheng Injection (the main ingredients are Codonopsis and Astragalus) in the treatment of digestive tract diseases were studied. Investigators found that Astragalus can not only inhibit the growth of pancreatic tumors, but also down regulate the ability of CAFs to secrete βig-h3, thereby inducing CD8+T proliferation and inhibiting the polarization of macrophages into M2 macrophages, thereby enhancing the response of pancreatic tumors to gemcitabine and other treatment options.

Thus, the objective of this study is to compare the impact of combining Astragalus with Gemcitabine versus Gemcitabine alone as neoadjuvant treatment for pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of pancreatic ductal adenocarcinoma;
* Is 18 years of age or older;
* ECOG performance status 0 to 2;

Patient organ function tests must meet the following laboratory parameters:

* Transaminases AST (SGOT) and ALT (SGPT) ≤ 2.5 times the upper limit of normal (ULN). If liver function abnormalities are due to underlying liver metastasis, then AST (SGOT) and ALT (SGPT) may be ≤ 5 times ULN.
* Total serum bilirubin ≤ 3.0 times ULN (if due to underlying liver metastasis, then total bilirubin may be ≤ 5 times ULN),
* Neutrophils 1,500/Ul,
* hemoglobin > 8.0 gm/dL,
* Platelet count ≥ 100,000/mm3 (IU: ≥ 100 x 109/L),
* serum creatinine < 2.0 mg/dL,
* Expected postoperative survival ≥ 3 months;
* Ability to comply with the study visit plan and other protocol requirements;
* Voluntary participation and signing of informed consent.
* Is willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* CNS damage or soft meningeal disease;
* Metastasis to distant sites;
* Other serious diseases or conditions, including congestive heart failure (New York Heart Association class III or IV), unstable angina pectoris, infarction in the past 6 months, severe arrhythmia, prolonged QT interval, active HIV infection or HIV disease, mental disorders, and substance abuse;
* Known hypersensitivity to Astragalus or gemcitabine;
* Pregnant or lactating women. Women of childbearing potential who are unwilling or unable to use an acceptable method of contraception throughout the treatment period of this trial and for 12 weeks after the last dose of study drug. Sexually active, fertile men who are not using effective contraception themselves if their partner is a woman of childbearing potential;
* Known neuroendocrine tumor of the pancreas;
* Receiving a concomitant treatment with drugs interacting with gemcitabine;
* Past or concurrent cancers with primary foci or histology completely different from pancreatic cancer, except for cervical cancer in situ, previously treated basal cell carcinoma, and superficial bladder tumors (Ta, Tis & T1). Any cancer cured >5 years prior to enrollment is allowed;
* Inability to swallow herbal medicines or untreated malabsorption syndrome and unwillingness to take herbal medicines.
* Patients with poor compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | From first dose of study medication until approximately 3 years
  Objective response rate (ORR) measures the overall treatment response by assessing the percentage of patients with complete or partial tumor shrinkage after treatment.

SECONDARY OUTCOMES:
Surgical resection rate | From first dose of study medication until approximately 1 year
  Surgical resection rate refers to the percentage of patients who undergo surgical removal (resection) of a tumor or diseased tissue as part of their medical treatment.
Percentage of patients with a 50% decrease in CA19-9 | From first dose of study medication until approximately 3 years
  Percentage of patients with a 50% decrease in CA19-9 measures the proportion of individuals whose CA19-9 tumor marker levels have reduced by at least 50%, indicating a potential positive response to treatment
Safety and Tolerance of Chemotherapeutic Drugs (CTCAE) | From first dose of study medication until 30 days after the end of treatment, up to approximately 3 years
  Safety and Tolerance of Chemotherapeutic Drugs refers to the assessment of adverse events and side effects associated with chemotherapy, using the Common Terminology Criteria for Adverse Events (CTCAE) scale, which evaluates the safety profile and tolerability of chemotherapy in patients.
Progression-free survival(PFS) | From first dose of study medication until disease progression, permanent discontinuation of study treatment, or death due to any cause, up to approximately 3 years
  From first dose of study medication until disease progression, permanent discontinuation of study treatment, or death due to any cause, up to approximately 3 years.
Overall Survival (OS) | From first dose of study medication until disease progression, permanent discontinuation of study treatment, or death due to any cause, up to approximately 3 years
  OS will be calculated as date of death minus date of first dose of study medication plus 1. In the absence of death confirmation, OS will be censored at the date of last study follow-up. Analysis will be performed by Kaplan-Meier method.
Proportion of participants with R0 resection | From first dose of study medication until approximately 1 year
  R0 resection rate signifies the percentage of surgical procedures in which the entire tumor is successfully removed with no residual cancerous tissue remaining (complete microscopic tumor removal).

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen University General Hospital, Shenzhen, Guangdong, China